CLINICAL TRIAL: NCT00569010
Title: Randomized Phase I/II Study of 5-Azacytidine in Combination With Cytosine Arabinoside in Patients With Relapsed/Refractory Acute Myelogenous Leukemia or High Risk Myelodysplastic Syndrome - "SPORE"
Brief Title: Phase I/II Study of 5-Azacytidine With Ara-C in Patients With Relapsed/Refractory Acute Myelogenous Leukemia (AML) or High Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0291
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Leukemia
Keywords: Acute Myelogenous Leukemia; AML; Myelodysplastic Syndrome; MDS; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia | interventions — Azacitidine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low-Dose Ara-C + AZA-Level 0 (Experimental): Group 1 = Low-Dose Ara-C + Azacitidine-Level 0
  Low-Dose Ara-C: 100 mg/m^2 Daily continuous intravenous infusion (CIV) for 7 days Azacitidine (AZA): 37.5 mg/m^2 intravenous (IV) Over 20-30 minutes Daily for 7 Days
  Interventions: Drug: Azacitidine; Drug: Ara-C
- Low-Dose Ara-C + AZA-Level 1 (Experimental): Group 2 = Low-Dose Ara-C + Azacitidine-Level 1
  Low-Dose Ara-C: 100 mg/m^2 Daily continuous intravenous infusion (CIV) for 7 days AZA: Level 1 = 75.0 mg/m^2 IV Over 20-30 minutes Daily for 7 days
  Interventions: Drug: Azacitidine; Drug: Ara-C
- High-Dose Ara-C + AZA-Level 0 (Experimental): Group 3 = High-Dose Ara-C + Azacitidine-Level 0 High-dose Ara-C: 1 g/m^2 Daily CIV for 4 days (age<65years) or 3 days (age>=65years) AZA: 37.5 mg/m^2 IV Over 20-30 minutes Daily for 7 Days
  Interventions: Drug: Azacitidine; Drug: Ara-C
- High-Dose Ara-C + AZA-Level 1 (Experimental): Group 4 = High-Dose Ara-C + Azacitidine-Level 1
  High-dose Ara-C: 1 g/m^2 Daily CIV for 4 days (age<65years) or 3 days (age>=65 years) AZA:Level 1 = 75.0 mg/m^2 IV Over 20-30 minutes Daily for 7 days
  Interventions: Drug: Azacitidine; Drug: Ara-C

INTERVENTIONS:
Drug: Azacitidine — Group 1 and 3 at Level 0 = 37.5 mg/m^2 IV Over 20-30 minutes Daily for 7 Days Group 2 and 4 at Level 1 = 75.0 mg/m^2 IV Over 20-30 minutes Daily for 7 days
  Other Names: Vidaza
Drug: Ara-C — Group 1 and 2 at Low-Dose = 100 mg/m^2 Daily continuous intravenous infusion (CIV) for 7 days
  Arms 3 and 4 at High-dose = 1 g/m^2 Daily CIV for 4 days (age<65 years) or 3 days (age>=65 years)
  Other Names: Cytosar-U; cytarabine; cytosine Arabinoside

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Azacytidine (5-azacytidine) combined with cytosine arabinoside (ara-C) for the treatment of patients with relapsed and/or refractory Acute Myeloid Leukemia (AML) or high-risk Myelodysplastic Syndrome (MDS). The safety and effectiveness of this treatment combination will also be studied.

DETAILED DESCRIPTION:
5-azacytidine is designed to "turn off" the growth of cancer cells. This may be increased by ara-C, which is designed to kills leukemia cells by helping to stop the cells from dividing.

If you are found to be eligible to take part in this study, you will be assigned to a treatment group. You will be randomly assigned (as in the toss of a coin) to one of the 4 treatment groups. The first 3 to 6 patients will be assigned to Group 1. If no serious side effects are experienced, the next 3 to 6 patients will be assigned to Group 2. If no serious side effects are experienced, the next 3 to 6 patients will be assigned to Group 3. If no serious side effects are experienced, the next 3 to 6 patients will be assigned to Group 4.

If you are in Group 1, you will receive low-dose 5-azacytidine as an infusion by vein over 20 to 30 minutes every day for 7 days. You will also receive low-dose ara-C as a continuous infusion by vein for 7 days.

If you are in Group 2, you will receive high-dose 5-azacytidine as an infusion by vein over 20 to 30 minutes every day for 7 days. You will also receive low-dose ara-C as a continuous infusion by vein for 7 days.

If you are in Group 3, you will receive low-dose 5-azacytidine as an infusion by vein over 20 to 30 minutes every day for 7 days. You will also receive high-dose ara-C as a continuous infusion by vein for 3 days (if you are 65 years of age or older) or for 4 days (if you are younger than 65 years of age).

If you are in Group 4, you will receive high-dose 5-azacytidine as an infusion by vein over 20 to 30 minutes every day for 7 days. You will also receive high-dose ara-C as a continuous infusion by vein for 3 days (if you are 65 years of age or older) or for 4 days (if you are younger than 65 years of age).

Each group's treatment will be repeated every 4 to 8 weeks (this is considered 1 cycle of treatment), depending on your blood counts and how well your bone marrow is recovering. You will receive at least 2 cycles of treatment. You will continue to receive treatment, unless your disease gets worse or if you experience intolerable side effects. If your disease gets worse or you experience intolerable side effects, you may be taken off this study.

This is an investigational study. 5-azacytidine has been approved by the FDA for the treatment of MDS. Ara-C has been approved by the FDA for the treatment of AML. Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed Acute Myeloid Leukemia (AML) or high risk and previously treated Myelodysplastic Syndrome (MDS).
2. Patients with (1) refractory disease or (2) first relapse within 6 months of therapy or (3) 2nd or more of relapse of Acute Myelogenous Leukemia (AML) or high risk Myelodysplastic Syndrome MDS will be considered for the study.
3. Patients must have been off chemotherapy for 4 weeks prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease.
4. Age >=18 years. Deoxyribonucleic acid (DNA) methylation plays a significant role in development, and the effects of azacitidine in children are not well described.
5. Patients must have normal organ as defined: Total bilirubin <2 mg, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) <2.5 x institutional upper limit of normal, Creatinine <2 mg
6. Ability to understand and the willingness to sign a written informed consent document.
7. Women of child bearing potential must have a negative serum pregnancy test prior to azacitidine treatment.
8. Women of child bearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with azacytidine.
9. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier, unless there is evidence of rapidly progressive disease. Patients may have received hydroxyurea prior to entering the study.
2. Patients may not be receiving any other investigational agents for their leukemias.
3. Patients with active brain or meningeal disease should be excluded.
4. Known or suspected hypersensitivity to azacitidine or mannitol
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
6. Pregnant women are excluded from this study because azacitidine is a Deoxyribonucleic acid (DNA) methyltransferase inhibitor which has teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with azacitidine, breastfeeding should be discontinued if the mother is treated with azacitidine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre Issa, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period 12/28/2005 to 8/25/2008. All participants were registered at The University of Texas M.D. Anderson Cancer Center.
Pre-assignment Details: Of the 36 enrolled, only 34 evaluable participants were included in this study and started study drug.
Groups:
- Low-Dose Ara-C + AZA-Level 0: Low-Dose Ara-C: 100 mg/m^2 Daily continuous intravenous infusion (CIV) for 7 days; Azacitidine (AZA): 37.5 mg/m^2 intravenous (IV) Over 20-30 minutes Daily for 7 Days
- Low-Dose Ara-C + AZA-Level 1: Low-Dose Ara-C: 100 mg/m^2 Daily continuous intravenous infusion (CIV) for 7 days AZA: Level 1 = 75.0 mg/m^2 IV Over 20-30 minutes Daily for 7 days
- High-Dose Ara-C + AZA-Level 0: Ara-C: 1 g/m^2 Daily CIV for 4 days (age<65years) or 3 days (age>=65years); AZA: 37.5 mg/m^2 IV Over 20-30 minutes Daily for 7 Days
- High-Dose Ara-C + AZA-Level 1: High-dose Ara-C: 1 g/m^2 Daily CIV for 4 days (age<65years) or 3 days (age>=65 years); AZA: Level 1 = 75.0 mg/m^2 IV Over 20-30 minutes Daily for 7 days
Period: Overall Study
Arm/Group | Low-Dose Ara-C + AZA-Level 0 | Low-Dose Ara-C + AZA-Level 1 | High-Dose Ara-C + AZA-Level 0 | High-Dose Ara-C + AZA-Level 1
Started | 6 | 6 | 11 | 11
Completed | 6 | 6 | 11 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Dose Ara-C + AZA-Level 0 | Low-Dose Ara-C + AZA-Level 1 | High-Dose Ara-C + AZA-Level 0 | High-Dose Ara-C + AZA-Level 1 | Total
Number analyzed (Participants) | 6 | 6 | 11 | 11 | 34
Age Continuous [Mean (Full Range); unit: years] | 44 [31 to 76] | 61 [49 to 75] | 74 [52 to 79] | 62 [38 to 69] | 61 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 5 | 15
  Male | 3 | 2 | 8 | 6 | 19
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 11 | 11 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Remission
Description: Clinical response is determined by achievement of a complete remission (CR) as judged by morphological criteria (< 1% blasts in bone marrow with neutrophil recovery) according to International Working Group (IWG) criteria.
Time Frame: 6 weeks
Population: Analysis was per protocol.
Measure: Number; unit: participants
Arm/Group | Low-Dose Ara-C + AZA-Level 0 | Low-Dose Ara-C + AZA-Level 1 | High-Dose Ara-C + AZA-Level 0 | High-Dose Ara-C + AZA-Level 1
Number analyzed (Participants) | 6 | 6 | 11 | 11
participants | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: 2 years 4 months
Arm/Group | Low-Dose Ara-C + AZA-Level 0 | Low-Dose Ara-C + AZA-Level 1 | High-Dose Ara-C + AZA-Level 0 | High-Dose Ara-C + AZA-Level 1
Serious Adverse Events (participants affected / at risk) | 5/6 | 5/6 | 8/11 | 3/11
Other Adverse Events (participants affected / at risk) | 3/6 | 0/6 | 0/11 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Ara-C + AZA-Level 0 (N=6) | Low-Dose Ara-C + AZA-Level 1 (N=6) | High-Dose Ara-C + AZA-Level 0 (N=11) | High-Dose Ara-C + AZA-Level 1 (N=11)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) — Unrelated to study drug
colotis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to study drug
Disease Progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to study drug
Heart Disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Intracranial Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) — Unrelated to study drug
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug
Cardiac Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug.
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Unrelated to study drug.
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Occular/Visual other 20/400 (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to study drug
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-Dose Ara-C + AZA-Level 0 (N=6) | Low-Dose Ara-C + AZA-Level 1 (N=6) | High-Dose Ara-C + AZA-Level 0 (N=11) | High-Dose Ara-C + AZA-Level 1 (N=11)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 5 (5)
Mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes